CLINICAL TRIAL: NCT06477341
Title: The Effect of Active Nutritional Support On The Incidence Of Mucositis And Quality Of Life In Patients With Head And Neck Cancer Receiving Radiotherapy
Brief Title: The Effect of Active Nutritional Support On Quality Of Life In Patients With Head And Neck Cancer Receiving Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Mohamed Aboelela Hassan, resident doctor at oncology department of Assiut university hospital, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RMAHassan
Record Dates: First submitted 2024-03-26; First posted 2024-06-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): patients of head and neck cancer receiving radiotherapy , who did not receive any nutritional support during radiotherapy
- nutritional support grouped (Active Comparator): patients of head and neck cancer receiving radiotherapy , who receive any nutritional support during radiotherapy whether oral or intravenous like dipeptivine for mucositis
  Interventions: Dietary Supplement: various available nutrition as those contain high protein content as ensure milk

INTERVENTIONS:
Dietary Supplement: various available nutrition as those contain high protein content as ensure milk — note effect with usually prescribed suitable oral and parenteral nutrition for head and neck cancers receiving radiotherapy
  Arms: nutritional support grouped

SUMMARY:
note effect of appropriate nutrition on head and neck cancer patients receiving radiotherapy

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the sixth most common cancer worldwide with more than half a million new cases diagnosed each year . Because of the limitations imposed by the complicated anatomical structure of the head and neck to the operation, radiotherapy (RT) has become the main treatment method for HNC. However, damage to the normal tissue surrounding the tumor is inevitable. The most common manifestations of injury caused by RT are mucositis with the dry mouth, loss of taste, and dysphagia. The severe dysphagia leads to a definitive total impossibility of eating through the mouth in 20-30% of patients. Radiation-induced oral mucositis (RIOM) is a common side effect after radiotherapy (RT) in head and neck cancer (HNC) patients. RIOM patients with severe pain have difficulty in eating, which increases the incidence of malnutrition and affects patients' quality of life and the process of RT.

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer patients with age >18
* Newly diagnosed head and neck cancer patients
* histological proven HNC cancer
* head and neck cancer patients treated with radiotherapy or chemo radiotherapy

Exclusion Criteria:

* Advanced and Metastatic head and neck cancer patients
* head and neck cancer patients treated with chemotherapy only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
nutritional status of patients | two years
  Follow up improvement by evaluating weight in kg and height in meters to calculate body mass index in kg / m^2

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdehtawab, lecturer, Study Chair — Assiut University
Locations (1):
- Reham mohamed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
when research is publicly puplished
Supporting Information: SAP
Time Frame: will be available after two years and used whenever it needed
Access Criteria: at scientific research magazines

REFERENCES:
- See also: Related Info — http://rehammohamed9891@gmail.com